CLINICAL TRIAL: NCT01847677
Title: A Randomized Phase II Multi-centric Open Label Clinical Trial to Determine the Efficacy and Toxicity of Preoperative Chemotherapy With or Without Bevacizumab in Patients With Advanced Ovarian Cancer
Brief Title: Neoadjuvant Therapy in Advanced Ovarian Cancer With Avastin
Acronym: NOVA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Investigación en Cáncer de Ovario (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEICO-1205; 2012-003883-31 (EudraCT Number)
Record Dates: First submitted 2013-04-26; First posted 2013-05-07 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2019-05

CONDITIONS: Cancer, Ovarian
Keywords: ovarian cancer; neoadyuvant; bevacizumab
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paclitaxel & Carboplatin (Active Comparator): 1. Preoperative treatment Cycle 1 to 4 (4 cycles every 3 weeks of chemotherapy pre-surgery)
     * Carboplatin AUC 6 i.v. first day
     * Paclitaxel 175 mg/m2 i.v. first day
  2. Surgery
  3. Post-Operative treatment
  Cycle 5 to 7 (3 cycles every 3 weeks of chemotherapy post-surgery):
  * Carboplatin AUC 6 i.v. first day
  * Paclitaxel 175 mg/m2 i.v. first day
  * Bevacizumab 15 mg/Kg i.v. first day1
  When the chemotherapy treatment is completed, the patient will continue with maintenance bevacizumab until 15 months length treatment.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin
- Paclitaxel & Carboplatin & Bevacizumab (Experimental): 4 cycles every 3 weeks (at least 3 Bevacizumab neoadjuvant cycles): Carboplatin AUC 6 i.v. first day Paclitaxel 175 mg/m2 i.v. first day Bevacizumab 15 mg/Kg i.v. first day.
  b) Surgery Ovarian cancer surgery should be performed according to FIGO guidelines.
  c) Postoperative treatment
  Both arms:
  Cycle 5 to 7 (3 cycles every 3 weeks of chemotherapy post-surgery):
  Carboplatin AUC 6 i.v. first day Paclitaxel 175 mg/m2 i.v. first day Bevacizumab 15 mg/Kg i.v. first day.
  When the chemotherapy treatment is completed, the patient will continue with maintenance bevacizumab until 15 months length treatment.
  Interventions: Drug: Bevacizumab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Bevacizumab
  Other Names: Avastin
  Arms: Paclitaxel & Carboplatin & Bevacizumab
Drug: Paclitaxel
  Other Names: Taxol
Drug: Carboplatin
  Other Names: Paraplatin

SUMMARY:
Recently results have shown that Bevacizumab is active both in monotherapy and in combination therapy in patients with ovarian cancer. One of our objectives is to evaluate whether the addition of neoadjuvant bevacizumab improves the response and whether this affects the evolution of patients.

DETAILED DESCRIPTION:
Epithelial ovarian cancer (OC) is the fourth leading cause of cancer death in women, after lung, breast and colon cancer, and it represents the most common cause of death from gynaecological malignancies. The high mortality associated with OC is due to the lack of screening tests that enable an early diagnosis, thus the majority of patients are diagnosed at advanced stages of the disease when the chances of a cure are very limited. In fact, the 5-year overall survival (OS) rate for stage III-IV OC does not exceed 20-30% in many series. The standard treatment for advanced OC is maximal cytoreductive surgery (or debulking) followed by the administration of 6 cycles of adjuvant chemotherapy with carboplatin and paclitaxel.

In recent years, a number of studies have been carried out with antiangiogenic drugs. Specifically, bevacizumab, an anti-VEGF monoclonal antibody, has been shown to be active both in monotherapy and combination therapy in patients with OC that have received multiple previous lines of chemotherapy.

One of the objectives is to evaluate whether the addition of neoadjuvant bevacizumab improves the response and whether this affects the evolution of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Women over 18 years old
2. Obtained informed consent, in writing and signed
3. Histological confirmation of primary peritoneal carcinoma or fallopian tube carcinoma
4. Planned interval debulking surgery
5. ECOG:0 to 2
6. Life expectancy >12 weeks

Exclusion Criteria:

1. Non-epithelial ovarian cancer, including malignant mixed Müllerian tumors.
2. Borderline ovarian tumors.
3. Administration of intraperitoneal chemotherapy planned.
4. Previous systemic anti-tumor treatment against ovarian cancer.
5. Intestinal obstruction or sub-occlusion, intestinal infiltration shown by CT scan or rectosigmoid infiltration in gynaecological examination.
6. Uncontrolled hypertension.
7. Any previous radiotherapy: abdomen or pelvis.
8. Major traumatic injuries in the 4 weeks prior to the first potential dose of bevacizumab.
9. History or clinical suspicion of brain metastases or spinal cord compression.
10. History or evidence of central nervous system (CNS) disorders, unless properly treated with standard medical treatment.
11. Cerebrovascular accident (CVA), transient ischemic attack (TIA) or subarachnoid haemorrhage (SAH) in the 6 months prior to randomization.
12. Fertile women of childbearing age who are not willing to use effective contraception during the study and at least 6 months after the study.
13. Women that are breastfeeding or pregnant.
14. Prior exposure to mouse CA-125 antibody.
15. Treatment with any other experimental product, or participation in another clinical trial within 30 days prior to inclusion.
16. Malignant tumors other than ovarian cancer within the 5 years prior to randomisation, with the exception of cervical carcinoma in situ treated correctly and/or basal-cell carcinoma.
17. Known hypersensitivity to bevacizumab or any of its excipients (including Cremophor).
18. Non-healing wound, active peptic ulcer or bone fracture. Patients with healing incised granulomas by secondary intention, with no evidence of fascial dehiscence or infection can be included, but they require three weeks of wound control.
19. History or evidence of bleeding or thrombotic diathesis
20. Current or recent continued use of aspirin > 325 mg / day (within 10 days prior to randomization)
21. Current or recent use (within 10 days before the first cycle of treatment) of full doses of anticoagulants or thrombolytics administered orally or parenterally for therapeutic purposes (except for vascular permeability, in which case the INR should be kept below 1.5).
22. Clinically significant cardiovascular disease, including:

    * Myocardial infarction or unstable angina (≤ 6 months before randomization)
    * Congestive heart failure (CHF) class ≥ II of the NYHA (New York Heart Association)
    * Poorly controlled cardiac arrhythmia despite medication (may include patients with atrial fibrillation with controlled frequency)
    * Peripheral vascular disease ≥ grade 3 (i.e. symptomatic and interfering with activities or daily living [ADL] needing repair or review)
23. Pre-existing sensory or motor neuropathy, ≥ grade 2
24. Demonstration of any other neurological or metabolic dysfunction involving a reasonable suspicion of the existence of a disease or condition that contraindicates the use of an experimental drug, or that involves an increased risk to the patient of treatment-related complications
25. No medical or psychiatric illness that may impede the performance of a systemic or surgical treatment
26. Laboratory:

Inadequate bone marrow function:

* ANC: <1.5 x 109/l
* platelet count <100 x 109/l
* Hb <9 g/dl. (Patients may be transfused)

Inadequate coagulation parameters: Activated partial thromboplastin time (APTT) >1.5 x ULN or INR >1.5

Inadequate liver function, defined as:

* Serum (total) bilirubin >1.5 x the upper limit of normal (ULN) for the institution
* AST & ALT > 2.5 x ULN (> 5 x ULN in patients with liver metastases) or alkaline phosphatase > 2.5 x ULN (or > 5 x ULN in case of liver metastases or > 10 x ULN in case of bone metastases).

Inadequate renal function, defined as:

* Serum creatinine >2.0 mg/dl or >177 mol/l
* Urine dipstick for proteinuria >2+
* Patients with 2+ proteinuria on baseline dipstick analysis should undergo a 24-hour urine collection and must demonstrate ≤1g of protein in their 24-hour urine collection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2013-05-06 (Actual); Primary Completion 2015-06-04 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Complete response rate | average 24 months
  Complete response rate (microscopic residual tumor included) assessed by the surgeon at laparotomy after neoadjuvant therapy.

SECONDARY OUTCOMES:
Safety: toxicities and surgical complications | average 24 months
  Safety and tolerability of the treatment will be assessed by adverse event description: incidence, severity, time of onset, causes, and abnormal laboratory values .
Surgical feasibility | average 24 months
  rate of patients in which surgery is feasible, comparing both arms.
Optimal surgery rate | average 24 months
  rate of patients in which surgery is optimal (residual disease<1cm), comparing both arms
RECIST 1.1 responses and correlation with serological responses (GCIG criteria) | average 24 months
  It will be assesed using descriptive statistics techniques such as frequency tables and contingency tables
Progression-free survival according RECIST 1.1 criteria | average 24 months
  tables of survival will be constructed by the Kaplan-Meier method. Mean and median, both with confidence intervals of 95%. Comparisons between groups will be made by log-rank test.
Overall Survival (OS) | average 24 months
  tables of survival will be constructed by the Kaplan-Meier method. Mean and median, both with confidence intervals of 95%. Comparisons between groups will be made by log-rank test.
Association between clinical response and the expression of protein biomarkers, in pre-and post-surgical plasma. | average 24 months
  It will be assesed using descriptive statistics techniques such as frequency tables and contingency tables
Biomarkers: Epithelial-mesenchymal transition performed at C.S. Parc Taulí | average 24 months
  It will be assesed using descriptive statistics techniques such as frequency tables and contingency tables

OTHER OUTCOMES:
Histological response: comparison between the obtained response only with chemotherapy or chemotherapy and bevacizumab. | average 24 months
  information correlating the clinical laboratory with the response to treatment.
Association of clinical response with other potential biomarkers, including but not limited to, single nucleotide polymorphisms (SNP) and specific tumor markers. | Average 24 months
  It will be assesed using descriptive statistics techniques such as frequency tables and contingency tables

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda García, MD, Study Chair — C.S Parc Taulí
Locations (13):
- Spain (13):
  - Hospital La Fe, Valencia, Valencia
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Clínic, Barcelona
  - Hospital Sant Pau, Barcelona
  - H. Reina Sofia, Córdoba
  - ICO Girona, Girona
  - ICO Hospitalet, Hospitalet Del Llobregat
  - Hospital 12 de Octubre, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Morales Meseguer, Murcia
  - Hospital Son Llatzer, Palma Mallorca
  - Parc Taulí, Sabadell
  - Hospital Marqués de Valdecilla, Santander

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961